CLINICAL TRIAL: NCT06164093
Title: Follow-up Study of Autologous Transplantation of P63+ Lung Progenitor Cells for Treatment of Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, Jieming QU, Principal Investigator, Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023318
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; P63+ lung progenitor cells; Autologous transplantation; Mechanism study
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects once received LPCs transplantation treatment (Other): The patients who have participated in the clinical trial of autologous transplantation of P63+ LPCs for treatment of bronchiectasis, and actually received LPCs transplantation treatment. (n = 15)
  Interventions: Other: RNA sequencing is performed on the remaining LPCs
- Subjects providing samples of surgically resected bronchiectasis lesions (Other): The bronchiectasis patients who could provide samples of surgically resected lung lesions. (n = 5)
  Interventions: Other: Immunofluorescence staining is performed in the surgically resected lung tissue sections

INTERVENTIONS:
Other: RNA sequencing is performed on the remaining LPCs — RNA sequencing is performed on the remaining LPCs previously transplanted back into the patients. And the results are analysed combined with the data from the previous clinical trial. (Please note that patients will not receive cell transplantation again as they have already received the treatment in the previous trial [NCT03655808])
  Arms: Subjects once received LPCs transplantation treatment
Other: Immunofluorescence staining is performed in the surgically resected lung tissue sections — The aim of this intervention is to detect Krt5 protein expression by staining the surgically resected lung tissue sections. This is done to confirm the presence of a small number of LPCs in the lung tissue of patients with bronchiectasis and to investigate their distribution.
  Arms: Subjects providing samples of surgically resected bronchiectasis lesions

SUMMARY:
This is the follow-up study of autologous transplantation of P63+ lung progenitor cells (LPCs) for treatment of bronchiectasis (NCT03655808). Bronchiectasis is the consequence of chronic suppurative inflammation and fibrosis of the bronchial tubes and the surrounding lung tissues. This seriously damages the muscular and elastic tissues of the bronchial walls, leading to deformation and permanent dilatation of the bronchial tubes. Histopathological damage to the patient's lungs is irremediable. However, there is no effective drug for rebuilding the damaged lung tissue structure, and thus cannot fully restore normal lung function. Lung progenitor cells, located in the basal position of the bronchial epithelium, express the P63 and Keratin-5 (KRT5) marker genes. These cells are active in division and migration, continuously generating new cells to replace other types of dead epithelial cells. They exhibit functional plasticity and can directly repair bronchial and alveolar structures. P63+ LPCs can be extracted by fibreoptic brushing and then isolated, purified and expanded on a large scale using appropriate methods. Currently, preclinical studies and some pilot clinical trials have shown that these cells can successfully repair damaged lungs, improve lung function and have a favourable safety profile. To further investigate the therapeutic mechanism of P63+ LPCs, RNA sequencing will be performed on the remaining LPCs previously transplanted back into the patients. Additionally, to confirm the existence of LPCs in the lung tissue of bronchiectasis patients, the pathological sections of lung tissue samples from patients who had received surgical resection of the lesions, will be subjected to fluorescence staining.

ELIGIBILITY:
Subjects once received cell treatment

Inclusion Criteria:

* Subjects diagnosed as bronchiectasis.
* Subjects have participated in the clinical trial of autologous transplantation of P63+ LPCs for treatment of bronchiectasis, and actually received LPCs transplantation treatment.
* Subjects with stable condition for more than 2 weeks.
* Subjects can tolerate bronchoscopy.
* Subjects signed informed consent.
* Subjects with good compliance.

Exclusion Criteria:

* Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
* Subjects with positive serological tests for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or syphilis (HBV carriers and patients with stable chronic hepatitis B could be accepted if titers of HBV DNA < 500 IU/mL or copies < 1000 copies/mL; patients with curative hepatitis C were eligible if HCV RNA tests were negative).
* Subjects with any malignancy.
* Subjects with any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, acute exacerbation of chronic bronchitis or extremely severe chronic obstructive pulmonary disease (COPD).
* Subjects with other serious diseases, such as diabetes, myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
* Subjects with leukopenia (WBC less than 4x10^9 / L) or agranulocytosis (WBC less than 1.5x10^9 / L or neutrophils less than 0.5x10^9 / L) caused by any reason.
* Subjects with severe renal impairment, serum creatinine> 1.5 times of the upper limit of normal.
* Subjects with liver disease or liver damage: alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin> 2 times of the upper limit of normal.
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
* Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
* Subjects with a history of alcohol or illicit drug abuse.
* Subjects accepted by any other clinical trials within 3 months before the enrollment.
* Subjects with poor compliance, difficult to complete the study.
* Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Subjects providing samples of surgically resected bronchiectasis lesions

Inclusion Criteria:

* Subjects diagnosed as bronchiectasis.
* Subjects have never participated in the clinical trial of autologous transplantation of P63+ LPCs for treatment of bronchiectasis, and never received LPCs transplantation treatment.
* Subjects have once received surgery to remove bronchiectasis lesions and lung samples are still kept in the Department of Pathology, Ruijin Hospital till now.
* Subjects signed informed consent.

Exclusion Criteria:

* Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
* Subjects with positive serological tests for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or syphilis (HBV carriers and patients with stable chronic hepatitis B could be accepted if titers of HBV DNA < 500 IU/mL or copies < 1000 copies/mL; patients with curative hepatitis C were eligible if HCV RNA tests were negative).
* Subjects with any malignancy.
* Subjects with any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, acute exacerbation of chronic bronchitis or extremely severe COPD.
* Subjects with a history of alcohol or illicit drug abuse.
* Subjects accepted by any other clinical trials within 3 months before the enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Different transcriptomic profiles of LPCs among the patients once received cell transplantation treatment | From date of inclusion until the date of final quantification, assessed up to 6 months
  RNA sequencing of remaining LPCs previously transplanted back into patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No